CLINICAL TRIAL: NCT02095795
Title: Effectiveness of an Exoskeleton Gait Training Versus Manual Therapy in Subacute Post Stroke Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Giovanni Taveggia (Other)
Responsible Party: Sponsor-Investigator, Giovanni Taveggia, Medical Director, Habilita, Ospedale di Sarnico
Organization: Habilita, Ospedale di Sarnico (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Habilita-RAR-05
Record Dates: First submitted 2014-02-27; First posted 2014-03-26 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Stroke
Keywords: Exercise Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Technological Rehabilitation (Experimental): Patients in the experimental group received a multimodal treatment intervention consisting of 60 minutes of conventional treatment according to the Bobath approach (Bobath B. Adult hemiplegia: evaluation and treatment. Oxford: Butterworth-Heineman, 1990) followed by 30 minutes of robotic gait training on the Lokomat robotic system with the supervision of an expert rehabilitator. Patients started the first session with 50% weight unload and 1.5 Km/h gait speed, performances increments are allowed only in the following sessions. Each patient received 20 sessions over a period of 4 weeks (5 sessions per week).
  Interventions: Device: Technological Rehabilitation
- Control Rehabilitation (Active Comparator): Patients in the control group received the same number of treatment sessions of a similar duration as those in the experimental group but they received activities of overground walking exercises targeted to improve walking in substitution of the robotic gait trainer.
  Interventions: Other: Control Rehabilitation

INTERVENTIONS:
Device: Technological Rehabilitation — The Lokomat (Hocoma, Zurich, Switzerland) is robotic device conformed as an exoskeleton on the lower limbs of the patient. Through active and passive actuators, it realize a proper trajectory with an associated motion profile of the involved limbs. The results are physically guide repetitive, rhythmic, bilateral lower extremity movements in order to simulate a physiological gait cycle.The system uses a dynamic body weight-support system to support the participant above a motorized treadmill synchronized with the Lokomat. Participants were provided verbal encouragement to actively step in conjunction with the movement presented by the Lokomat.
  Other Names: Lokomat
  Arms: Technological Rehabilitation
Other: Control Rehabilitation — When needed, more than one therapist are employed in the intervention for safety reasons.
  Other Names: Manual rehabilitation with the therapist.
  Arms: Control Rehabilitation

SUMMARY:
The main objective of the present study was to compare the effects of exoskeleton devices used in electromechanical-assisted gait training after stroke compared to over ground conventional physical therapy in a single blind research.

The second objective is to research when the devices can be used with the best chance of success in the functional recovery of gait in people who are unable to walk independently after stroke.

DETAILED DESCRIPTION:
Stroke is the leading cause of death and of serious long term disability in adults, three mouths after stroke, 20% of people remain wheelchair bound, and 70% walk at reduced velocity and capacity.

People who suffer a stroke, when regain ambulatory function, walk with typically asymmetrical gait pattern, slow, and metabolically inefficient. These characteristics are associated with difficulty advancing and bearing weight though the more affected limb, leading to instability and increased risk of falls.

Manually-assisted body-weight supported Treadmill training (BWSTT) is a contemporary approach to gait rehabilitation after stroke, whereas an individual walks on a treadmill, the therapists manually facilitate hemiparetic limb and trunk control in an effort to normalize upright reciprocal stepping and dynamic postural control. Advantages of this approach are that little to no ambulatory function is required to initiate locomotion and early post stroke training effects are transferred of improvements in over ground gait including: symmetry, speed, and endurance as well as motor impairment and balance scores.

An example of electromechanical devices is Lokomat, a robotic gait orthosis combined with harness-supported body weight system is used together with a treadmill. However the main difference from treadmill training is that the patient's legs are guided by the robotic device according to a preprogrammed gait pattern. A computer-controlled robotic gait orthosis guides the patient, and the process of gait training in automated.

Lokomat can be used to give non ambulatory patients intensive practice in terms of high repetitions, of complex gait cycles with a reduced effort for therapists, as they no longer need to set the paretic limbs or assist trunk movements.

The main objective of the present study was to compare the effects of exoskeleton devices used in electromechanical-assisted gait training after stroke compared to over ground conventional physical therapy in a single blind research.

The second objective is to research when the devices can be used with the best chance of success in the functional recovery of gait in people who are unable to walk independently after stroke.

ELIGIBILITY:
Inclusion Criteria:

* hemiparesis at least six months from stroke.

Exclusion Criteria:

* Ashworth scale >3
* Bone instability (unconsolidated fractures, vertebral instability, severe osteoporosis),
* Articular ankyloses, contractures
* Spasms with locomotion effects
* Mini Mental State Examination (MMSE) [???] < 22 points and behavioral diseases involving aggressivity or psychotic disorders
* Clinicopathological conditions contraindicating the rehabilitation treatment (respiratory insufficiency, cardiac/circulatory failure, osteomyelitis, phlebitis and other conditions)
* Cutaneous lesions at lower limbs
* Weight > 135 kg
* Height > 200 cm
* Dysmetria of lower limbs more than 2 cm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Gait performances | 1 day before the treatment
  All evaluation procedures are performed by the same examiner who was blinded to the aims of the study and to which group the participants are allocated.
  The 6-Minute Walk Test (6MWT) and 10 meters walking test are used to assess endurance and speed, respectively. The 6MWT quantifies functional mobility based on the distance in meters traveled in 6 minutes. This outcome is a measure of endurance and is particularly significant to evaluate the possibility to perform continuative tasks, that are particularly important for the rehabilitation of stroke patients and are relevant for an autonomous life.
  The speed is quantified with the 10-meters Walk Test (TWT) over the ground. The gait speed measurement is performed over the middle six meters of the TWT and patients are asked to walk at their comfortable speed.
Gait performances | 1 day after the treatment
  All evaluation procedures are performed by the same examiner who was blinded to the aims of the study and to which group the participants are allocated.
  The 6-Minute Walk Test (6MWT) and 10 meters walking test are used to assess endurance and speed, respectively. The 6MWT quantifies functional mobility based on the distance in meters traveled in 6 minutes. This outcome is a measure of endurance and is particularly significant to evaluate the possibility to perform continuative tasks, that are particularly important for the rehabilitation of stroke patients and are relevant for an autonomous life.
  The speed is quantified with the 10-meters Walk Test (TWT) over the ground. The gait speed measurement is performed over the middle six meters of the TWT and patients are asked to walk at their comfortable speed.
Gait performances | 60 days after the treatment
  All evaluation procedures are performed by the same examiner who was blinded to the aims of the study and to which group the participants are allocated.
  The 6-Minute Walk Test (6MWT) and 10 meters walking test are used to assess endurance and speed, respectively. The 6MWT quantifies functional mobility based on the distance in meters traveled in 6 minutes. This outcome is a measure of endurance and is particularly significant to evaluate the possibility to perform continuative tasks, that are particularly important for the rehabilitation of stroke patients and are relevant for an autonomous life.
  The speed is quantified with the 10-meters Walk Test (TWT) over the ground. The gait speed measurement is performed over the middle six meters of the TWT and patients are asked to walk at their comfortable speed.

SECONDARY OUTCOMES:
Functional outcomes | 1 day before the treatment
  Functional Ambulation Category (FAC)
Functional outcomes | 1 day before the treatment
  Ashworth Scale
Functional outcomes | 1 day before the treatment
  Functional Independence Measure (FIM)
Functional outcomes | 1 day before the treatment
  Motricity Index Right
Functional outcomes | 1 day before the treatment
  Motricity Index Left
Functional outcomes | 1 day before the treatment
  National Institute of Health Stroke Scale (NIHSS)
Functional outcomes | 1 day before the treatment
  Numerical Rating Pain Scale
Functional outcomes | 1 day before the treatment
  Quality of Life (SF36)
Functional outcomes | 1 day before the treatment
  Tinetti Gait Test
Functional outcomes | 1 day before the treatment
  Tinetti Balance Test
Functional outcomes | 1 day after the treatment
  Functional Ambulation Category (FAC)
Functional outcomes | 60 days after the treatment
  Functional Ambulation Category (FAC)
Functional outcomes | 1 day after the treatment
  Ashworth Scale
Functional outcomes | 60 days after the treatment
  Ashworth Scale
Functional outcomes | 1 day after the treatment
  Functional Independence Measure (FIM)
Functional outcomes | 60 days after the treatment
  Functional Independence Measure (FIM)
Functional outcomes | 1 day after the treatment
  Motricity Index Right
Functional outcomes | 60 days after the treatment
  Motricity Index Right
Functional outcomes | 1 day after the treatment
  Motricity Index Left
Functional outcomes | 60 days after the treatment
  Motricity Index Left
Functional outcomes | 1 day after the treatment
  National Institute of Health Stroke Scale (NIHSS)
Functional outcomes | 60 days after the treatment
  National Institute of Health Stroke Scale (NIHSS)
Functional outcomes | 1 day after the treatment
  Numerical Rating Pain Scale
Functional outcomes | 60 days after the treatment
  Numerical Rating Pain Scale
Functional outcomes | 1 day after the treatment
  Quality of Life (SF36)
Functional outcomes | 60 days after the treatment
  Quality of Life (SF36)
Functional outcomes | 1 day after the treatment
  Tinetti Gait Test
Functional outcomes | 60 days after the treatment
  Tinetti Gait Test
Functional outcomes | 1 day after the treatment
  Tinetti Balance Test
Functional outcomes | 60 days after the treatment
  Tinetti Balance Test

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Taveggia, Physician, Principal Investigator — Habilita, Ospedale di Sarnico
Locations (2):
- Italy (2):
  - Habilta Zingonia, Ciserano, BG
  - Habilita Sarnico, Sarnico, BG